CLINICAL TRIAL: NCT00327418
Title: A Double Blind Placebo Controlled Study of Atorvastatin as Prevention of CHD in High Risk Patients With Non-Insulin Dependent Diabetes Mellitus (Collaborative Atorvastatin Study - CARDS)
Brief Title: CARDS Is Designed To Show If Lowering Cholesterol With Atorvastatin In Type 2 Diabetics Without CV Disease Reduces The Risk Of CV Events
Acronym: CARDS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Diabetes UK (Other); Department of Health, United Kingdom (Other Government)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 0981-430-102; A2581143
Record Dates: First submitted 2006-05-16; First posted 2006-05-18 (Estimated); Last update posted 2007-05-10 (Estimated); Status verified 2007-05

CONDITIONS: Major Coronary Event; Cerebrovascular Accident; Coronary Artery Bypass Graft; Angina, Unstable; Revascularization
MeSH Terms: conditions — Stroke; Angina, Unstable | interventions — Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin

SUMMARY:
A study to assess the efficacy of once daily atorvastatin 10 mg versus placebo on cardiovascular endpoints in patients with non-insulin-dependent diabetes mellitus (NIDDM) who have a history of either hypertension, retinopathy, microalbuminuria, macroalbuminuria, or who currently smoke, but who do not have established corornary heart disease or other macrovascular disease.

ELIGIBILITY:
Inclusion Criteria:

Patients must have a documented history of at least one of the following:

* Hypertension (defined as systolic blood pressure 140 mmHg or a diastolic blood pressure 90 mmHg (defined as the disapperance of all sound [Korotkoff Phase V] or receiving anti-hypertensive treatment. Blood pressure should be measured after sitting the patient quietly for 3 minutes).
* Retinopathy (defined as any of the following; non-proliferative retinopathy, pre-pre-proliferative retinopathy, proliferative retinopathy, maculopathy, advanced diabetic eye disease or history of photocoagulation).
* Microalbuminuria (defined as either, Albumin creatinine ratio > than = to 2.5 mg/mmol, or Albumin excretion rate on a timed collection > than = to 20 mcg/min (> than = to 30 mg/24hrs) on two successive occasions, or a positive micral or other strip test).
* Macroalbuminuria (defined as either; Albustix or other dipstick evidence of gross proteinuria, Albumin creatinine ratio > than = to 25 mg/mmol; or Albumin excretion rate on a timed collection > than = 200 mcg/min (> than = 300 mg/24hrs) on two sucessive occasions).
* Current smoker

Exclusion Criteria:

* Type I Diabetes Mellitus
* Any major Coronary event prior to entry into the study

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2800
Dates: Start 1997-01; Study Completion 2004-02

PRIMARY OUTCOMES:
Time from randomization to the occurrence of a primary clinical endpoint
i.e. major coronary event or CABG or other coronary revascularization procedure
or unstable angina or resuscitated cardiac arrest or stroke.

SECONDARY OUTCOMES:
The incidence rate of a primary clinical and endpoint; the time from randomization
to the occurrence of and the incidence rate of other parameters e.g. total
mortality, any cardiovascular event, new PVD etc. and the percent change from
baseline in various lipid and lipoprotein parameters.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (107):
- United Kingdom (107):
  - Pfizer Investigational Site, Fosterhill, Aberdeen
  - Pfizer Investigational Site, Irvine, Ayrshire
  - Pfizer Investigational Site, Midsomer Norton, Bath
  - Pfizer Investigational Site, Reading, Berkshire
  - Pfizer Investigational Site, Slough, Berkshire
  - Pfizer Investigational Site, Maidenhead, Berskhire
  - Pfizer Investigational Site, Edgbaston, Birmingham
  - Pfizer Investigational Site, Frenchay, Bristol
  - Pfizer Investigational Site, Llanishen, Cardiff
  - Pfizer Investigational Site, Wrexham, Clwydd
  - Pfizer Investigational Site, Bocastle, Cornwall
  - Pfizer Investigational Site, Falmouth, Cornwall
  - Pfizer Investigational Site, Fowey, Cornwall
  - Pfizer Investigational Site, Penzance, CORNWALL
  - Pfizer Investigational Site, Penzance, Cornwall
  - Pfizer Investigational Site, Redruth, Cornwall
  - Pfizer Investigational Site, Saltash, CORNWALL
  - Pfizer Investigational Site, St Austell, Cornwall
  - Pfizer Investigational Site, Truro, Cornwall
  - Pfizer Investigational Site, Chesterfield, Derbyshire
  - Pfizer Investigational Site, Crownhill, Plymouth, DEVON
  - Pfizer Investigational Site, Plymouth, Devon
  - Pfizer Investigational Site, Plympton, Devon
  - Pfizer Investigational Site, Bournemouth, Dorset
  - Pfizer Investigational Site, Epping, Essex
  - Pfizer Investigational Site, Southend-on-Sea, Essex
  - Pfizer Investigational Site, Langside, Glasgow
  - Pfizer Investigational Site, Portsmouth, Hampshire
  - Pfizer Investigational Site, Southampton, Hampshire
  - Pfizer Investigational Site, Titchfield, Hampshire
  - Pfizer Investigational Site, Hemel Hempstead, Hertfordshire
  - Pfizer Investigational Site, Watford, Hertfordshire
  - Pfizer Investigational Site, Ryde, Isle of Wight
  - Pfizer Investigational Site, Gillingham, Kent
  - Pfizer Investigational Site, Hildenborough, Kent
  - Pfizer Investigational Site, Royal Tunbridge Wells, Kent
  - Pfizer Investigational Site, Bolton, Lancashire
  - Pfizer Investigational Site, Ormskirk, Lancashire
  - Pfizer Investigational Site, Waterloo, Liverpool
  - Pfizer Investigational Site, Manchester, M15 6SX
  - Pfizer Investigational Site, Ashford, Middlesex
  - Pfizer Investigational Site, Southall, Middlesex
  - Pfizer Investigational Site, Scunthorpe, North Lincolnshire
  - Pfizer Investigational Site, Harrogate, North Yorkshire
  - Pfizer Investigational Site, Northallerton, North Yorkshire
  - Pfizer Investigational Site, Sutton in Ashfield, Nottinghamshire
  - Pfizer Investigational Site, Worksop, Nottinghamshire
  - Pfizer Investigational Site, Huthwaite, Nottingham
  - Pfizer Investigational Site, Headington, Oxford
  - Pfizer Investigational Site, Haverfordwest, Pembrokeshire
  - Pfizer Investigational Site, Shrewsbury, Shropshire
  - Pfizer Investigational Site, Frome, Somerset
  - Pfizer Investigational Site, Weston-super-Mare, Somerset
  - Pfizer Investigational Site, Sheffield, South Yorkshire
  - Pfizer Investigational Site, Stirling, Stirlingshire
  - Pfizer Investigational Site, Carshalton, Surrey
  - Pfizer Investigational Site, Epsom, Surrey
  - Pfizer Investigational Site, Pontarddulais, Swansea
  - Pfizer Investigational Site, Dundee, Tayside
  - Pfizer Investigational Site, Hetton-Le-Hole, Tyne & Wear
  - Pfizer Investigational Site, Gateshead, Tyne and Wear
  - Pfizer Investigational Site, Nuneaton, Warwickshire
  - Pfizer Investigational Site, Rugby, Warwickshire
  - Pfizer Investigational Site, Lyndon, West Bromwich, West Midlands
  - Pfizer Investigational Site, Livingston, West Lothian
  - Pfizer Investigational Site, Wolverhampton, West Midlands
  - Pfizer Investigational Site, Crawley, West Sussex
  - Pfizer Investigational Site, Haywards Heath, West Sussex
  - Pfizer Investigational Site, Corsham, Wiltshire
  - Pfizer Investigational Site, Trowbridge, Wiltshire
  - Pfizer Investigational Site, Warminster, Wiltshire
  - Pfizer Investigational Site, Westbury, Wiltshire
  - Pfizer Investigational Site, York, Yorkshire
  - Pfizer Investigational Site, Ayr
  - Pfizer Investigational Site, Bath
  - Pfizer Investigational Site, Belfast
  - Pfizer Investigational Site, Birmingham
  - Pfizer Investigational Site, Cambridge
  - Pfizer Investigational Site, Chippenham, Wiltshire
  - Pfizer Investigational Site, Co. Dublin
  - Pfizer Investigational Site, Coventry
  - Pfizer Investigational Site, Derby
  - Pfizer Investigational Site, Dewsbury
  - Pfizer Investigational Site, Dublin
  - Pfizer Investigational Site, Dumfries
  - Pfizer Investigational Site, East Kilbride
  - Pfizer Investigational Site, Edinburgh
  - Pfizer Investigational Site, Glasgow
  - Pfizer Investigational Site, Hartlepool
  - Pfizer Investigational Site, Hertfordshire
  - Pfizer Investigational Site, Inverness
  - Pfizer Investigational Site, Leicester
  - Pfizer Investigational Site, Liverpool
  - Pfizer Investigational Site, Llantrisant
  - Pfizer Investigational Site, London
  - Pfizer Investigational Site, Manchester
  - Pfizer Investigational Site, Newcastle upon Tyne
  - Pfizer Investigational Site, Nottingham
  - Pfizer Investigational Site, Oldham
  - Pfizer Investigational Site, Paisley
  - Pfizer Investigational Site, Pontefract
  - Pfizer Investigational Site, Southampton
  - Pfizer Investigational Site, Swansea
  - Pfizer Investigational Site, Wakefield
  - Pfizer Investigational Site, Wigan
  - Pfizer Investigational Site, Wiltshire
  - Pfizer Investigational Site, Wishaw

REFERENCES:
- [Result] Neil HA, DeMicco DA, Luo D, Betteridge DJ, Colhoun HM, Durrington PN, Livingstone SJ, Fuller JH, Hitman GA; CARDS Study Investigators. Analysis of efficacy and safety in patients aged 65-75 years at randomization: Collaborative Atorvastatin Diabetes Study (CARDS). Diabetes Care. 2006 Nov;29(11):2378-84. doi: 10.2337/dc06-0872. PMID 17065671
- [Derived] Tunnicliffe DJ, Palmer SC, Cashmore BA, Saglimbene VM, Krishnasamy R, Lambert K, Johnson DW, Craig JC, Strippoli GF. HMG CoA reductase inhibitors (statins) for people with chronic kidney disease not requiring dialysis. Cochrane Database Syst Rev. 2023 Nov 29;11(11):CD007784. doi: 10.1002/14651858.CD007784.pub3. PMID 38018702
- [Derived] Vogt L, Bangalore S, Fayyad R, Melamed S, Hovingh GK, DeMicco DA, Waters DD. Atorvastatin Has a Dose-Dependent Beneficial Effect on Kidney Function and Associated Cardiovascular Outcomes: Post Hoc Analysis of 6 Double-Blind Randomized Controlled Trials. J Am Heart Assoc. 2019 May 7;8(9):e010827. doi: 10.1161/JAHA.118.010827. PMID 31020900
- [Derived] Bangalore S, Fayyad R, DeMicco DA, Colhoun HM, Waters DD. Body Weight Variability and Cardiovascular Outcomes in Patients With Type 2 Diabetes Mellitus. Circ Cardiovasc Qual Outcomes. 2018 Nov;11(11):e004724. doi: 10.1161/CIRCOUTCOMES.118.004724. PMID 30571333
- [Derived] Ports WC, Fayyad R, DeMicco DA, Laskey R, Wolk R. Effectiveness of Lipid-Lowering Statin Therapy in Patients With and Without Psoriasis. Clin Drug Investig. 2017 Aug;37(8):775-785. doi: 10.1007/s40261-017-0533-0. PMID 28573499
- [Derived] Deedwania PC, Pedersen TR, DeMicco DA, Breazna A, Betteridge DJ, Hitman GA, Durrington P, Neil A; TNT, CARDS and IDEAL Steering Committees and Investigators. Differing predictive relationships between baseline LDL-C, systolic blood pressure, and cardiovascular outcomes. Int J Cardiol. 2016 Nov 1;222:548-556. doi: 10.1016/j.ijcard.2016.07.201. Epub 2016 Jul 30. PMID 27513651
- [Derived] Kaasenbrood L, Poulter NR, Sever PS, Colhoun HM, Livingstone SJ, Boekholdt SM, Pressel SL, Davis BR, van der Graaf Y, Visseren FL; CARDS, ALLHAT, and ASCOT Investigators. Development and Validation of a Model to Predict Absolute Vascular Risk Reduction by Moderate-Intensity Statin Therapy in Individual Patients With Type 2 Diabetes Mellitus: The Anglo Scandinavian Cardiac Outcomes Trial, Antihypertensive and Lipid-Lowering Treatment to Prevent Heart Attack Trial, and Collaborative Atorvastatin Diabetes Study. Circ Cardiovasc Qual Outcomes. 2016 May;9(3):213-21. doi: 10.1161/CIRCOUTCOMES.115.001980. Epub 2016 May 11. PMID 27174798
- [Derived] Soedamah-Muthu SS, Livingstone SJ, Charlton-Menys V, Betteridge DJ, Hitman GA, Neil HA, Bao W, DeMicco DA, Preston GM, Fuller JH, Stehouwer CD, Schalkwijk CG, Durrington PN, Colhoun HM; CARDS Investigators. Effect of atorvastatin on C-reactive protein and benefits for cardiovascular disease in patients with type 2 diabetes: analyses from the Collaborative Atorvastatin Diabetes Trial. Diabetologia. 2015 Jul;58(7):1494-502. doi: 10.1007/s00125-015-3586-8. Epub 2015 Apr 22. PMID 25899452
- [Derived] Deshmukh HA, Colhoun HM, Johnson T, McKeigue PM, Betteridge DJ, Durrington PN, Fuller JH, Livingstone S, Charlton-Menys V, Neil A, Poulter N, Sever P, Shields DC, Stanton AV, Chatterjee A, Hyde C, Calle RA, DeMicco DA, Trompet S, Postmus I, Ford I, Jukema JW, Caulfield M, Hitman GA. Genome-wide association study of genetic determinants of LDL-c response to atorvastatin therapy: importance of Lp(a). J Lipid Res. 2012 May;53(5):1000-1011. doi: 10.1194/jlr.P021113. Epub 2012 Feb 24. PMID 22368281
- [Derived] Colhoun HM, Betteridge DJ, Durrington PN, Hitman GA, Neil HA, Livingstone SJ, Charlton-Menys V, DeMicco DA, Fuller JH; CARDS Investigators. Effects of atorvastatin on kidney outcomes and cardiovascular disease in patients with diabetes: an analysis from the Collaborative Atorvastatin Diabetes Study (CARDS). Am J Kidney Dis. 2009 Nov;54(5):810-9. doi: 10.1053/j.ajkd.2009.03.022. Epub 2009 Jun 21. PMID 19540640
- [Derived] Charlton-Menys V, Betteridge DJ, Colhoun H, Fuller J, France M, Hitman GA, Livingstone SJ, Neil HA, Newman CB, Szarek M, DeMicco DA, Durrington PN. Apolipoproteins, cardiovascular risk and statin response in type 2 diabetes: the Collaborative Atorvastatin Diabetes Study (CARDS). Diabetologia. 2009 Feb;52(2):218-25. doi: 10.1007/s00125-008-1176-8. Epub 2008 Oct 30. PMID 18972097
- [Derived] Newman CB, Szarek M, Colhoun HM, Betteridge DJ, Durrington PN, Hitman GA, Neil HA, Demicco DA, Auster S, Fuller JH; Cards Investigators. The safety and tolerability of atorvastatin 10 mg in the Collaborative Atorvastatin Diabetes Study (CARDS). Diab Vasc Dis Res. 2008 Sep;5(3):177-83. doi: 10.3132/dvdr.2008.029. PMID 18777490
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=0981-430-102&StudyName=CARDS+is+designed+to+show+if+lowering+cholesterol+with+atorvastatin+in+Type+2+diabetics+without+CV+disease+reduces+